CLINICAL TRIAL: NCT04522323
Title: A Phase 1b, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Antitumor Activity of MEDI5752 in Combination With Axitinib in Subjects With Advanced Renal Cell Carcinoma
Brief Title: A Study to Evaluate MEDI5752 and Axitinib in Subjects With Advanced Renal Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7980C00003; 2023-509604-15-00 (Registry Identifier: CTIS); 2019-004338-41 (EudraCT Number)
Record Dates: First submitted 2020-07-22; First posted 2020-08-21 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Advanced Renal Cell Carcinoma
Keywords: renal cell carcinoma; MEDI5752; PD-1/CTLA-4 bispecific; PD-1; CTLA-4; bispecific; axitinib; lenvatinib
MeSH Terms: conditions — Carcinoma, Renal Cell; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Axitinib; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Exploration (Experimental): The Dose exploration Phase is made up of Part A, B and Part C. Part A will evaluate the safety and tolerability of MEDI5752 in combination with Axitinib (2 patients), and Part B and C will evaluate the safety and tolerability of MEDI5752 in combination with Lenvatinib (~72 patients)
  Interventions: Biological: MEDI5752; Drug: Axitinib; Drug: Lenvatinib
- Dose Expansion (Experimental): Evaluate safety and anti-tumor activity of MEDI5752 in combination with Lenvatinib (~105 patients )
  Interventions: Biological: MEDI5752; Drug: Axitinib; Drug: Lenvatinib

INTERVENTIONS:
Biological: MEDI5752 — MEDI5752
Drug: Axitinib — INLYTA
Drug: Lenvatinib — LENVIMA

SUMMARY:
The purpose of this study is to evaluate MEDI5752 in combination with Lenvatinib (or Axitinib), in subjects with advanced renal cell carcinoma.

DETAILED DESCRIPTION:
The purpose of this Phase 1b study is to evaluate the safety, tolerability, pharmacokinetics, immunogenicity, and antitumor activity of MEDI5752 in combination with Lenvatinib (or Axitinib) in subjects with advanced renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 at the time of screening
* Body weight > 35 kg
* Written informed consent
* Histologically or cytologically proven advanced RCC with clear cell component
* Advanced RCC not previously treated in that setting
* Provision of tumor material (≥ 5 unstained slides or tissue block) from an archival or fresh tissue sample
* ECOG performance status of 0 or 1
* Subjects must have at least 1 measurable lesion according to RECIST v1.1
* Life expectancy ≥ 12 weeks
* Adequate organ and marrow function
* Female subjects of childbearing potential must have negative pregnancy test at screening and prior to each administration of investigational product, and must use at least one highly effective method of contraception.
* Strongly recommend nonsterilized male partners of female subjects of childbearing potential use a male condom plus spermicide from screening to 7.6 months after the last dose of MEDI5752 and 30 days after the last dose of lenvatinib.

Exclusion Criteria:

* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results
* Concurrent enrollment in another clinical study, unless it is an observational study.
* Previous treatment with mTOR inhibitors, PD-1, PD-L1, or CTLA-4 inhibitors for RCC or any other immune checkpoint inhibitor
* Previous treatment with VEGF inhibitors
* Evidence of the following infections: active infection including tuberculosis, human immunodeficiency virus, chronic or active hepatitis B or chronic or active hepatitis C
* History of organ transplant
* Active or prior documented autoimmune or inflammatory disorders
* Current or prior use of immunosuppressive medication within 14 days prior to the first dose of investigational product.
* Poorly controlled blood pressure (BP) defined as systolic BP ≥ 140/90 mmHg at screening and not able to be controlled prior to Cycle 1 Day 1 and any change in antihypertensive medications within 1 week prior to Cycle 1 Day 1.
* Thromboembolic (arterial or venous) events within previous 6 months
* Any concurrent therapy for cancer
* Receipt of live attenuated vaccine within 30 days prior to the first dose of investigational product
* Known allergy or hypersensitivity to investigational product(s) or any of the excipients of the investigational product(s)
* Untreated or progressive CNS metastatic disease, any leptomeningeal disease, or cord compression
* History of another primary malignancy
* Unresolved toxicities from previous anticancer therapy
* Major surgery within 4 weeks prior to enrollment or radiation therapy within 2 weeks prior to enrollment or has not recovered from AEs due to prior treatment
* Female subjects must not breastfeed and must not donate, or retrieve for their own use, ova from screening to 3 months after the last dose of MEDI5752 and 30 days after the last dose of lenvatinib.
* History of arrhythmia which is symptomatic or requires treatment, symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia
* Uncontrolled intercurrent illness within the last 6 months prior to enrollment
* Clinically significant gastrointestinal abnormality
* Serious nonhealing wound, ulcer, or bone fracture
* Has clinically significant hemoptysis (at least 0.5 teaspoon of bright red blood) or tumor bleeding within 2 weeks before the first dose of investigational product
* Radiographic evidence of major blood vessel invasion/infiltration/encasement

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2025-09-26 (Estimated); Study Completion 2025-09-26 (Estimated)

PRIMARY OUTCOMES:
Number of subjects experiencing adverse events (AEs)/serious adverse events (SAEs) | Informed consent through 90-Day Post Last Dose.
  The primary safety endpoint is as assessed by the number of subjects with adverse events and serious adverse events (SAEs) graded per NCI CTCAE v5.0.
Number of Participants With Dose Limiting Toxicities (DLT) of MEDI5752 and Lenvatinib (or Axitinib) during the Dose Exploration period. | Informed consent through the first 21 days of treatment with MEDI5752 and Lenvatinib (or Axitinib) in the Dose Exploration Period.
  Determine the MTD and recommended Phase 2 dose (RP2D) of the combination of MEDI5752 and Lenvatinib.
  A dose limiting toxicity (DLT) is defined as MEDI5752 treatment-related AE of any Grade 3 or higher toxicity (as defined in the protocol) CTCAE v5.0.
Number of subjects experiencing adverse events (AEs) leading to discontinuation. | Informed consent through 90-Day Post Last Dose.
  The primary safety endpoint is as assessed by the number of subjects with serious adverse events (SAEs) graded per NCI CTCAE v5.0.
Number of subjects experiencing abnormal laboratory evaluations. | Informed Consent through 90 post treatment date.
  The primary safety endpoint is as assessed by the number of subjects experiencing changes in laboratory evaluations from baseline.
Number of subjects experiencing changes in vital signs reported as Adverse Events. | Informed consent through 90-Day Post Last Dose
  The primary safety endpoint is assessed by the change in vital signs from baseline.
Number of subjects experiencing abnormal electrocardiograms (ECG) reported as Adverse Events. | Informed consent through 90-Day Post Last Dose
  The primary safety endpoint is as assessed by the change in ECG parameters from baseline.
Preliminary antitumor activity of MEDI5752 combined with Lenvatinib (or Axitinib) by Objective response rate per RECIST version (v) 1.1. | First subject enrolled through 18 months from last subject enrolled, an average of 30 months.
  The primary efficacy endpoint is assessed by the antitumor activity of MEDI5752 combined with Lenvatinib.

SECONDARY OUTCOMES:
Antitumor activity of MEDI5752 combined with Lenvatinib by measuring the progression free survival (PFS) according to RECIST v1.1. | Last Subject Enrolled through study completion, an average of 48 months.
  The endpoint for assessment of PFS is defined as the time from the first dose of treatment until the documentation of PD or death due to any cause, whichever occurs first.
Antitumor activity of MEDI5752 combined with Lenvatinib by measuring the Best Overall Response (BOR) according to RECIST v1.1. | First subject enrolled through 18 months from last subject enrolled, an average of 30 months.
  The endpoint for assessment of BOR will be based on all post-baseline disease assessments that occur prior to the initiation of subsequent anticancer treatment
Antitumor activity of MEDI5752 combined with Lenvatinib by measuring the Disease Control Rate (DCR). | Informed Consent through the date of first documented progression, end of study, date of death, or two years after last subject starts treatment whichever should occur first
  The endpoint for assessment of DCR is measured by the proportion of subjects with a BOR of confirmed CR, PR, or SD.
Antitumor activity of MEDI5752 combined with Lenvatinib by measuring the Duration of Response (DOR) according to RECIST v1.1. | Informed Consent through the date of first documented progression, end of study, date of death, or two years after last subject starts treatment whichever should occur first
  The endpoint for assessment of DOR is measured by the duration from the first documented OR to the first documented PD or death due to any cause, whichever occurs first.
Antitumor activity of MEDI5752 combined with Lenvatinib by measuring the Time to Response (TTR) according to RECIST v1.1. | Informed Consent through the date of first documented progression, end of study, date of death, or two years after last subject starts treatment whichever should occur first
  The endpoint for assessment of TTR is defined as the time from the first dose of treatment until the first documentation of an OR.
Pharmacokinetics of MEDI5752: Cmax | Day 1, 8, 15, 22, 64 and then Day 1 of every other cycle
  The endpoints for the assessment of PK of MEDI5752 include individual MEDI5752 concentrations at different time points after administration.
Pharmacokinetics of MEDI5752: AUC | Day 1, 8, 15, 22, 64 and then Day 1 of every other cycle
  The endpoints for the assessment of PK of MEDI5752 include individual MEDI5752 concentrations at different time points after administration.
Pharmacokinetics of MEDI5752: Cmin | Day 1, 8, 15, 22, 64 and then Day 1 of every other cycle
  The endpoints for the assessment of PK of MEDI5752 include individual MEDI5752 concentrations at different time points after administration.
Pharmacokinetics of MEDI5752: t 1/2 | Day 1, 8, 15, 22, 64 and then Day 1 of every other cycle
  The endpoints for the assessment of PK of MEDI5752 include individual MEDI5752 concentrations at different time points after administration.
Pharmacokinetics of MEDI5752: Clearance | Day 1, 8, 15, 22, 64 and then Day 1 of every other cycle
  The endpoints for the assessment of PK of MEDI5752 include individual MEDI5752 concentrations at different time points after administration.
Immunogencity of MEDI572: Incidence of ADAs against MEDI5752 | Day 1, 8, 15, 22, 30, 64 and then Day 1 of every other cycle
  The endpoints for the immunogenicity of MEDI5752 include the number of subjects who develop detectable anti-drug antibodies (ADAs) to MEDI5752.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Early Oncology, Study Director — AstraZeneca
Locations (16):
- United States (7):
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Fort Myers, Florida
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Hershey, Pennsylvania
  - Research Site, Nashville, Tennessee
- Australia (2):
  - Research Site, Frankston
  - Research Site, Waratah
- Research Site, Villejuif, France
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Sabadell
  - Research Site, Seville
  - Research Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home